CLINICAL TRIAL: NCT00446277
Title: Corneal Endothelial Cell Loss in Diabetes Type II During Cataract Surgery
Status: Suspended | Type: Observational
Why Stopped: The present study was joining 2005-41-4933 into one study
Sponsor: Frederiksberg University Hospital (Other)
Other Study IDs: ASP01
Record Dates: First submitted 2007-03-09; First posted 2007-03-12 (Estimated); Last update posted 2008-05-12 (Estimated); Status verified 2008-05

CONDITIONS: Diabetes Mellitus
Keywords: cataract surgery, endothelial cell, cell loss, diabetes; mellitus type II
MeSH Terms: conditions — Diabetes Mellitus | interventions — Cataract Extraction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: cataract surgery

SUMMARY:
The aim of the present study is to evaluate changes in the morphology and function of the corneal endothelium before and after cataract surgery in patients with diabetes type II. Also to explain if determination of HgbA1c in diabetics is a predictor for the changes in morphology and function.

DETAILED DESCRIPTION:
Thirty patients with Diabetes type II and thirty non-diabetes patients scheduled to cataract surgery (phacoemulsification with intraocular lens implantation) were invited to participate in the study. Preoperatively, all patients had a full eye examination and 3 endothelial cell photos were taken.

Three months postoperatively the patients were called for a re-examination including 3 endothelial cell photos. The function of the cornea is dependent of the number and morphology of the endothelial cells, and even small traumas like cataract surgery may disrupt the cornea integrity leading to corneal haze and blur. Diabetics may be more vulnerable to corneal stress.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cataract scheduled for surgery

Exclusion Criteria:

* Patients with corneal diseases, glaucoma or uveitis, previous intraocular surgery or eye traumas.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-01; Primary Completion 2007-06 (Estimated); Study Completion 2007-06 (Estimated)

PRIMARY OUTCOMES:
corneal endothelial cell count (cells / mm2)
percentage of hexagonal cells
variation in cell size
central corneal thickness

SECONDARY OUTCOMES:
visual acuity
intraocular pressure

CONTACTS AND LOCATIONS:
Overall Officials: Allan Storr-Paulsen, MD, Principal Investigator — Frederiksberg University Hospital
Locations (1):
- Department of Ophthalmology, Frederiksberg University Hospital, Frederiksberg, Copenhagen, Denmark